CLINICAL TRIAL: NCT03301597
Title: A Phase 2 Open-Label, Multi-Center, Randomized, Controlled, Dose-Finding Study of NLA101 in Adults Receiving High Dose Chemotherapy for Acute Myeloid Leukemia
Brief Title: NLA101 in Adults Receiving High Dose Chemotherapy for AML
Acronym: LAUNCH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development plan under review.
Sponsor: Nohla Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NLA-0101-CIN-01
Record Dates: First submitted 2017-09-27; First posted 2017-10-04 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Chemotherapy-induced Neutropenia; Bacterial Infections; Fungal Infections
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Bacterial Infections; Mycoses | interventions — Standard of Care; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to 1 of 3 Investigational Arms or a Control Arm in a 1:1:1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control Arm (Other): The Control Arm will receive standard of care (SOC) chemotherapy without the infusion of NLA101. SOC chemotherapy will be determined by local PI and must be a standard regimen for untreated de novo or secondary AML that will result in moderate to severe myelosuppression and will be given with curative intent.
  Interventions: Drug: Standard of Care (SOC) chemotherapy
- Low Dose Arm (Experimental): The Low Dose Arm will receive standard of care (SOC) chemotherapy with the infusion of low-dose NLA101.
  Interventions: Biological: NLA101; Drug: Standard of Care (SOC) chemotherapy
- Medium Dose Arm (Experimental): The Medium Dose Arm will receive standard of care (SOC) chemotherapy with the infusion of medium-dose NLA101.
  Interventions: Biological: NLA101; Drug: Standard of Care (SOC) chemotherapy
- High Dose Arm (Experimental): The High Dose Arm will receive standard of care (SOC) chemotherapy with the infusion of high-dose NLA101.
  Interventions: Biological: NLA101; Drug: Standard of Care (SOC) chemotherapy

INTERVENTIONS:
Biological: NLA101 — NLA101 is a universal donor "off-the-shelf" ex-vivo expanded hematopoietic stem and progenitor cell (HSPC) product that is cryopreserved and ready for immediate use.
  Other Names: Dilanubicel
  Arms: High Dose Arm; Low Dose Arm; Medium Dose Arm
Drug: Standard of Care (SOC) chemotherapy — The SOC chemotherapy regimen for each patient will be determined by local PI. Regimen must be a standard AML regimen that will result in moderate to severe myelosuppression and have curative intent.

SUMMARY:
Phase 2 open-label, multi-center, randomized, controlled, dose-finding study of safety and efficacy of NLA101 to reduce the rate of infections associated with CIN in adult subjects with AML.

DETAILED DESCRIPTION:
Phase 2 open-label, multi-center, randomized, controlled, dose-finding study of safety and efficacy of NLA101 to reduce the rate of infections associated with chemotherapy induced neutropenia (CIN) in adult subjects with AML.

Eligible subjects with untreated de novo or secondary AML and per local institutional standards planned to receive at least two cycles of chemotherapy with curative intent will be enrolled into the study and randomized 1:1:1:1 to 1 of 3 Investigational Arms (Standard of Care [SOC] chemotherapy + low, medium, or high dose NLA101) or a Control Arm (SOC chemotherapy).

Subjects randomized to an Investigational Arm will be eligible to receive a single fixed assigned dose of NLA101 after the first cycle of chemotherapy, and up to 2 additional identical cell doses after subsequent chemotherapy cycles (one NLA101 infusion per cycle). Subjects randomized to the Control Arm will be followed for up to 3 cycles of chemotherapy.

All subjects will be followed for 84 days following randomization, or 30 days post final infusion of NLA101, or 30 days post the day after the last chemotherapy infusion for Control Arm, whichever is longer.

ELIGIBILITY:
Key Criteria:

Inclusion Criteria:

* Age ≥ 18 (or legal age of majority for sites outside US).
* Untreated de novo or secondary acute myeloid leukemia (AML), including AML that has progressed from myelodysplastic syndrome (MDS), and histologically documented diagnosis
* Eligible for at least 2 cycles of standard of care AML chemotherapy that will result in moderate to severe myelosuppression and have curative intent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2 or Karnofsky Status of 50 to 100.
* Adequate cardiac, renal, and hepatic functions.

Exclusion Criteria:

* Extramedullary disease in the absence of bone marrow or blood involvement
* Acute promyelocytic leukemia (APL) with PML-RARA
* Prior AML therapy, with the exception of intrathecal chemotherapy or emergent radiation for myeloid sarcoma.
* Concurrent malignancy requiring active treatment with chemotherapy, immunotherapy, or radiation
* Prior allotransplant, including allogeneic hematopoietic cell transplant or solid organ allogeneic transplant
* Known hypersensitivity or history of hypersensitivity to dimethylsulfoxide (DMSO)
* Active/chronic human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Recurrent Event Rate of Grade 3 or Higher Bacterial or Fungal Infection | From randomization through follow-up of 84 days post randomization, 30 days post last infusion of NLA101, or 30 days post last infusion of chemotherapy for Control Arm, whichever is later

SECONDARY OUTCOMES:
Event rate of grade 3 or higher documented bacterial and fungal infections per cycle of chemotherapy | From randomization through follow-up of 84 days post randomization, 30 days post last infusion of NLA101, or 30 days post last infusion of chemotherapy for Control Arm, whichever is later
Incidence and duration of filgrastim (or biosimilar) administration | From randomization through follow-up of 84 days post randomization, 30 days post last infusion of NLA101, or 30 days post last infusion of chemotherapy for Control Arm, whichever is later
Overall Response Rate | From randomization through follow-up of 84 days post randomization, 30 days post last infusion of NLA101, or 30 days post last infusion of chemotherapy for Control Arm, whichever is later
Incidence and duration of complications due to infections | From randomization through follow-up of 84 days post randomization, 30 days post last infusion of NLA101, or 30 days post last infusion of chemotherapy for Control Arm, whichever is later
Incidence and duration of febrile neutropenia | From randomization through follow-up of 84 days post randomization, 30 days post last infusion of NLA101, or 30 days post last infusion of chemotherapy for Control Arm, whichever is later

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Tallman, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Naval G Daver, MD, Study Chair — M.D. Anderson Cancer Center
Locations (36):
- United States (25):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center - Fred & Pamela Buffett Cancer Center, Omaha, Nebraska
  - Westchester Medical Center, Hawthorne, New York
  - Weill Cornell Medical College - NewYork-Presbyterian Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai and Mount Sinai Health System, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Duke University Heath System, Duke Cancer Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert Hospital and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St. George Hospital, Kogarah, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Epworth HealthCare, Richmond, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- South Korea (4):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea's Seoul St. Mary's Hospital, Seoul